CLINICAL TRIAL: NCT02903576
Title: Stem Cell Derived Retinal Pigmented Epithelium Implantation in Patients With Outer Retinal Degenerations: Phase I/II Clinical Trial
Brief Title: Stem Cell Therapy for Outer Retinal Degenerations
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Rubens Belfort Jr., Full Professor of Ophthalmology, Federal University of São Paulo
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12018712.5.0000.5505
Record Dates: First submitted 2016-03-07; First posted 2016-09-16 (Estimated); Last update posted 2020-07-22 (Actual); Status verified 2017-08

CONDITIONS: Age Related Macular Degeneration; Stargardt's Disease; Exudative Age-related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration; Stargardt Disease | interventions — Suspensions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- injection of hESC-RPE in suspension (Active Comparator): 6 patients will receive cell suspension injections on the sub retinal space prior to the surgeries, to access safety
  Interventions: Procedure: injection of hESC-RPE in suspension
- injection hESC-RPE seeded in a substrate (Active Comparator): 15 patients will receive a sub-retinal implantation of a polymeric scaffold seeded hesc- RPE in monolayer
  Interventions: Procedure: injection hESC-RPE seeded in a substrate

INTERVENTIONS:
Procedure: injection of hESC-RPE in suspension — The first six patients will receive a sub retinal injection of hESC-RPE in solution after a complete pars plana vitrectomy to access safety of the cell implant alone.
  Other Names: Human Embryonic Stem Cell - Retinal Pigmented Epithelium
  Arms: injection of hESC-RPE in suspension
Procedure: injection hESC-RPE seeded in a substrate — Fifteen patients will receive a sub-retinal implantation of embryonic stem cell derived retinal pigmented epithelium seeded in a polymeric substrate to access safety of substrate seeded with RPE
  Other Names: Human Embryonic Stem Cell seeded in a polymeric substrate
  Arms: injection hESC-RPE seeded in a substrate

SUMMARY:
This study is a Phase I/II , open label,non randomized, prospective study to determine the safety of human embryonic stem cell derived Retinal pigmented epithelium (hESC RPE) sub retinal injections versus hESC RPE seeded on a polymeric substrate implanted in the sub retinal space,

DETAILED DESCRIPTION:
To determine whether the surgical implantation of a human embryonic stem cell-derived retinal pigmented epithelium (hESC-RPE) monolayer seeded onto a polymeric versus hESC-RPE injections into the sub retinal space is a safe procedure.

6 Patients will receive hESC-RPE cell injections (100000 cells) in the sub retinal space (2 Dry Age-related macular degeneration (AMD), 2 Wet AMD with disciform scar and 2 with Stargardt's disease).

Also 5 patients Dry AMD, 5 patients with Wet AMD with disciform scar and 5 patients with Stargardt's disease with receive a subretinal implantation of the hESC-RPE seeded in a monolayer in a polymeric substrate.

Patients will be enrolled sequentially, and after the procedure the patients will be followed for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients with AMD ( Dry , Wet after failure of treatment, disciform scars)
* Patients with Stargardt's Disease BCVA on the selected eye: worse than 20/200

Exclusion Criteria:

* Other ophthalmological diseases( Glaucoma, Diabetic Retinopathy, Previous retinal surgery, uveitis)
* Systemic diseases with contraindication for surgical procedures with local anaesthesia

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-08; Primary Completion 2019-01 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events of sub retinal implantation of stem cell derived retinal pigmented epithelium in the sub retinal space. | 1 year
  Incidence of surgical related side effects: Retinal detachment, Ocular inflammation, Increase in intraocular pressure, Infection( endophthalmitis), Loss of vision due to surgical, related complications

SECONDARY OUTCOMES:
Incidence of side effects related to the treatment itself( injection and implantation of sub retinal stem cell related RPE) | 1 year
  Inflammation/rejection Cell migration/differentiation Tumor formation Proliferative vitreoretinopathy/Retinal detachment Implant migration

CONTACTS AND LOCATIONS:
Overall Officials: Rubens Belfort, MD, Study Chair — Federal University of São Paulo UNIFESP
Locations (1):
- Federal University of Sao Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
scientific publication in a peer review journal